CLINICAL TRIAL: NCT01473472
Title: On Demand Antiretroviral Pre-exposure Prophylaxis for HIV Infection in Men Who Have Sex With Men
Acronym: IPERGAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-002645-35; IPERGAY (Other: ANRS)
Record Dates: First submitted 2011-11-08; First posted 2011-11-17 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection
Keywords: Prophylaxis; HIV infection; tenofovir; emtricitabine; men who have sex with men
MeSH Terms: conditions — HIV Infections; Homosexuality | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Truvada (Active Comparator): associated with an overall offer of prevention (counselling, STD screening, condoms, HAV and HBV vaccinations, treatment post-exposure to the HIV infection)
  Interventions: Drug: Truvada
- Placebo of Truvada (Placebo Comparator): associated with an overall offer of prevention (counselling, STD screening, condoms, HAV and HBV vaccinations, treatment post-exposure to the HIV infection)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Truvada — 2 tablets of truvada within 24 hours before first sexual relations, then 1 tablet of Truvada during the period of sexual activity including the last sexual intercourse, finally, a last dose of 1 tablet of Truvada approximately 24 hours later
  Other Names: tenofovir disoproxil and emtricitabine
  Arms: Truvada
Drug: Placebo — 2 tablets of placebo within 24 hours before first sexual relations, then 1 tablet of placebo every 24 hours during the period of sexual activity including the last sexual intercourse, finally, a last dose of 1 tablet of placebo approximatively 24 hours later
  Arms: Placebo of Truvada

SUMMARY:
This phase III, multi-centre, comparative, double-blind, randomized trial on 2 parallel groups is designed to evaluate a strategy for the prevention of HIV infection including "on demand" antiretroviral pre-exposure with Truvada versus placebo, associated with overall prevention (counselling, condoms, sexually transmitted diseases (STD) screening, hepatitis B virus (HBV) and hepatitis A virus (HAV) vaccinations and post-exposure treatment of HIV infection) in men who have sex with men (MSM), exposed to the risk of HIV infection. Indeed recent studies have reported a higher incidence of new HIV infection in MSM as compared to the general population, new approaches to the prevention of HIV infection are, therefore, necessary in order to consider the limits of current strategies.

DETAILED DESCRIPTION:
The trial has been taken place in two phases in order to ensure the general feasibility of the study:

* a first enrollment phase for at least 300 participants to ensure the possibility for recruitment in France and Canada and to validate the tools put into place as part of the trial to enroll and follow participants
* a second phase of 1600 additional participants. This extension phase started on July 2014.

The recruitment has been suspended following the recommendations of Data Safety and Monitoring Board (DSMB): the placebo arm has been stopped and Truvada was available for all the participants of the trial since November 2014. The initial protocol was amended and 361 participants were enrolled in the open-label phase. Sub-studies were proposed to the participants:

* Sub-study on the outcome of participants receiving sofosbuvir/ledipasvir treatment for recent HCV infection (protocol amendment on April 2015)
* Randomized sub-study to evaluate the efficacy of doxycycline post-exposure prophylaxis on sexually transmitted infections (protocol amendment on July 2015)
* Sub-study to evaluate Truvada adherence with Medication Event Monitoring System (MEMS) (protocol amendment on December 2015)
* Sub-study on drugs use and the impact on sexual behavior and Truvada adherence (protocol amendment on December 2015).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Male (or transgender) having sex with men
* Not infected with HIV-1 or HIV-2
* Elevated risk of HIV contamination : anal sexual relations with at least 2 different sexual partners within the past 6 months without the systematic use of a condom
* Satisfactory kidney function with a clearance of more than 60 mL/min (Cockcroft formula)
* Alanine aminotransferase (ALT) < 2.5 Upper Limit of Normal (ULN),
* Neutrophil granulocytes ≥ 1 000/mm3, haemoglobin ≥ 10 g/dL, platelets ≥ 150 000/mm3
* Negative HBs antigen and negative hepatitis C virus (HCV) serology (or negative HCV PCR if positive serology)
* Agrees to be contacted personally, if possible by telephone, short message system (SMS) or e-mail
* Agrees to the constraints imposed by the trial (visits every 2 months)
* Subjects enrolled in or a beneficiary of a Social Security program (State Medical Aid or Aide médicale de l'Etat (AME) is not a Social Security program).
* Signature of the informed consent form.

Exclusion Criteria:

* Subject in a stable and exclusive relationship with a person
* Systematic use of a condom during sexual relations
* Expected to go abroad for more than 3 consecutive months or move expected to a city where the study is not being conducted.
* Presence of significant glycosuria or proteinuria > 1+ in the urine dipstick, in the absence of infection.
* Presence of significant haematuria or leukocyturia > 2+ in the urine dipstick, in the absence of infection.
* History of chronic kidney disease, osteoporosis, osteopaenia
* History of pathological bone fracture not related to trauma
* Treatment with Interferon, Interleukin, or antiretrovirals
* Treatment that could inhibit or compete with the tubular secretion of antiretrovirals
* Treatment undergoing investigation
* Intravenous toxicomania
* Subject who is currently receiving or going to receive a potentially nephrotoxic treatment (long-term anti-inflammatory)
* Gastro-intestinal disease (or chronic nausea or vomiting) disrupting the absorption of treatments
* Positive HBs antigen
* Positive HCV serology with positive HCV PCR
* Life-threatening disease (lymphoma) or other serious disease (cardiovascular, renal, pulmonary, unstable diabetes) that could require treatment that could disrupt adherence to the treatment
* Subject potentially non-compliant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Contamination with HIV-1 or -2 | From randomization to the end of the trial. The trial end date will be set by the scientific committee when the necessary number of primary endpoints has been reached without exceeding 5 years of follow-up.
  The primary endpoint criteria is contamination with HIV-1 or -2, defined by the first diagnostic proof of infection: positive HIV serum test (using combined latest-generation tests HIV-1 + 2) or a positive test for HIV-1-RNA Polymerase Chain Reaction (PCR) in the plasma.

SECONDARY OUTCOMES:
Evolution of sexual behavior and potential at-risk behavior | Every 2 months without exceeding 5 years of follow-up.
  Self-questionnaires
Incidence of clinical and biological adverse events | From randomization to the end of the trial, without exceeding 5 years of follow-up.
Treatment adherence | Every 2 months without exceeding 5 years of follow-up.
  Self-questionnaires, pill count. Drugs levels in plasma and hair (every 4 months).
Incidence of hepatitis B | From randomization to the end of the trial, without exceeding 5 years of follow-up
Incidence of other sexually transmitted diseases | From randomization to the end of the trial, without exceeding 5 years of follow-up
Frequency of HIV resistance to antiretrovirals in HIV infected subjects | At a visit as soon as the HIV infection is diagnosed
  Genotype
Emtricitabine and tenofovir concentrations in plasma, saliva and rectal samples. | 0, 30 min, 1, 2, 4, 8 and 24 hours post-dose (2 tablets of Truvada)
  Ancillary study proposed between week-4 and the randomization - 12 volunteers. Blood and saliva samples at all time points and 2 sessions with rectal biopsies at two times for each volunteer (one before the drug is taken and one at one time after taking the 2 tablets)
Costs evaluation | From randomization to the end of the trial, without exceeding 5 years of follow-up.
  Modelling to estimate an increase of years of life expectancy and of quality adjusted life year (QALY).
  Cost per avoided HIV contamination

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel MOLINA, Professor, Principal Investigator — Hôpital Saint-Louis Paris FRANCE
Locations (7):
- CHUM - Hôpital Hôtel Dieu, Montreal, Canada
- France (6):
  - Hôpital de La Croix Rousse, Lyon
  - CHU Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Hôpital Gustave Dron, Tourcoing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chawki S, Leturque N, Minier M, Gabassi A, Foubert V, Charreau I, Cua E, Pialoux G, Meyer L, Molina JM, Delaugerre C. Prevalence and Risk Factors of Cytomegalovirus Among Men Having Sex With Men Enrolled in a Pre-Exposure Prophylaxis Study. Open Forum Infect Dis. 2024 Jul 18;11(8):ofae400. doi: 10.1093/ofid/ofae400. eCollection 2024 Aug. PMID 39100527
- [Derived] Antoni G, Tremblay C, Delaugerre C, Charreau I, Cua E, Rojas Castro D, Raffi F, Chas J, Huleux T, Spire B, Capitant C, Cotte L, Meyer L, Molina JM; ANRS IPERGAY study group. On-demand pre-exposure prophylaxis with tenofovir disoproxil fumarate plus emtricitabine among men who have sex with men with less frequent sexual intercourse: a post-hoc analysis of the ANRS IPERGAY trial. Lancet HIV. 2020 Feb;7(2):e113-e120. doi: 10.1016/S2352-3018(19)30341-8. Epub 2019 Nov 26. PMID 31784343
- [Derived] Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, Capitant C, Rojas-Castro D, Fonsart J, Bercot B, Bebear C, Cotte L, Robineau O, Raffi F, Charbonneau P, Aslan A, Chas J, Niedbalski L, Spire B, Sagaon-Teyssier L, Carette D, Mestre SL, Dore V, Meyer L; ANRS IPERGAY Study Group. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018 Mar;18(3):308-317. doi: 10.1016/S1473-3099(17)30725-9. Epub 2017 Dec 8. PMID 29229440
- [Derived] Molina JM, Charreau I, Spire B, Cotte L, Chas J, Capitant C, Tremblay C, Rojas-Castro D, Cua E, Pasquet A, Bernaud C, Pintado C, Delaugerre C, Sagaon-Teyssier L, Mestre SL, Chidiac C, Pialoux G, Ponscarme D, Fonsart J, Thompson D, Wainberg MA, Dore V, Meyer L; ANRS IPERGAY Study Group. Efficacy, safety, and effect on sexual behaviour of on-demand pre-exposure prophylaxis for HIV in men who have sex with men: an observational cohort study. Lancet HIV. 2017 Sep;4(9):e402-e410. doi: 10.1016/S2352-3018(17)30089-9. Epub 2017 Jul 23. PMID 28747274
- [Derived] Molina JM, Capitant C, Spire B, Pialoux G, Cotte L, Charreau I, Tremblay C, Le Gall JM, Cua E, Pasquet A, Raffi F, Pintado C, Chidiac C, Chas J, Charbonneau P, Delaugerre C, Suzan-Monti M, Loze B, Fonsart J, Peytavin G, Cheret A, Timsit J, Girard G, Lorente N, Preau M, Rooney JF, Wainberg MA, Thompson D, Rozenbaum W, Dore V, Marchand L, Simon MC, Etien N, Aboulker JP, Meyer L, Delfraissy JF; ANRS IPERGAY Study Group. On-Demand Preexposure Prophylaxis in Men at High Risk for HIV-1 Infection. N Engl J Med. 2015 Dec 3;373(23):2237-46. doi: 10.1056/NEJMoa1506273. Epub 2015 Dec 1. PMID 26624850
- See also: sponsor of the study — http://www.anrs.fr